CLINICAL TRIAL: NCT04094935
Title: Anterior Plate Osteosynthesis of Fractures of the Lower Extremity of the Radius: Does the Systematic Use of Short Epiphysic Screws Limit the Posterior Protrusion of the Screws Without Compromising Stability
Acronym: SHORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 190158; 2019-A00429-48 (Other: ANSM)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Fracture; Radius, Lower or Distal End
Keywords: Fracture of the radius
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anterior plate osteosynthesis of fractures of the lower extremity of the radius may be accompanied by tendinous complications : tenosynovitis of extensors or even tendon ruptures caused by the end of the epiphyseai screws.

The intraoperative measurements as well as the realization of the scopic pictures make it possible to estimate the length of the screws but the tendinous lesions remain frequent (5 to 15% according to the various series)

DETAILED DESCRIPTION:
* Preoperative consultation

  * Oral information of the patient of the protocol and delivery of the written information note
  * Seeking patient's non-opposition to participating in the study
  * Inclusion of the patient
* Surgical procedure for distal radius fracture + immediate post-operative radiography

  * Intervention performed according to the usual practices of the service by the surgeon of the day without randomization
  * Radiography: 2 shots: face and wrist profile
* Control X-ray + consultation

  * Achieved at 3 weeks, 6 weeks and 3 months after the intervention
  * X-rays: 2 shots: face and wrist profile
* Control ultrasound o Realized at 3 months after the intervention

End of participation in the study after consultation of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Fracture (s) of extra joint distal radius with or without joint refend in the sagitta plane
* Osteosynthesis by anterior locked plate
* Patient who did not oppose his participation in this research

Exclusion Criteria:

* Distal radius fractures with joint refend frontal (posterior marginal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients operated on for a fractured distal radius with an anterior locked plate in orthopaedic and trauma surgery in Saint Antoine Hospital, Paris
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Screws exceeding the posterior cortical | 3 months
  Proportion of tendon complications induced by conflict between the distal end of the epiphysal screws and extender tendons: rupture, tenosynovitis.

SECONDARY OUTCOMES:
Tendon complications | 3 months
  Proportion of tendon complications induced by conflict between the distal end of the epiphysal screws and extender tendons: rupture, tenosynovitis.
Secondary displacement or dismantling | 3 months
  Proportion of secondary displacement or dismantling 3-month control radio equipment (change of the radial slope on the face and radial glene's anversion on the profile between X-rays at J0 and control x-rays)
Ablation of material or resumption early surgery | 3 months
  Proportion of ablation of material or resumption early surgery on secondary displacement rated at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERISSON, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- St Antoine hospital - orthopaedic and traumatic surgery, Paris, France

IPD SHARING:
Plan to Share IPD: No